CLINICAL TRIAL: NCT02583568
Title: Phase II, Open-Label Study to Evaluate Safety and Explore Efficacy of Escalating Doses of Bevacizumab-IRDye800CW as an Optical Imaging Agent to Detect Cancer Tissue Delineation During Tumor Resection Surgery in Patients With Breast Cancer
Brief Title: Fluorescence Guided Surgery in Breast Cancer
Acronym: MARGIN
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Martini Hospital Groningen (Other)
Responsible Party: Principal Investigator, G.M. van Dam, prof.dr., University Medical Center Groningen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NL52447.042.15
Record Dates: First submitted 2015-06-30; First posted 2015-10-22 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Breast Cancer
Keywords: breast cancer; image-guided surgery
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Part 1 (Experimental): In part 1 a dose escalation will be performed for the tracer bevacizumab-800CW in four different dose groups (4,5mg 10mg 25mg 50mg)
  Interventions: Drug: Bevacizumab-800CW
- Part 2 (Experimental): In part 2, the two best performing dose groups of bevacizumab-800CW of part 1 will be expanded to a total of 10 patients per group.
  Interventions: Drug: Bevacizumab-800CW

INTERVENTIONS:
Drug: Bevacizumab-800CW — three days prior to surgery bevacizumab-800CW will be administered
  Other Names: Bevacizumab-IRDye800CW

SUMMARY:
A need for further investigation for fluorescence image-guided surgery in breast conserving surgery (BCS) has arisen following the results obtained from a phase I feasibility breast cancer trial (BIRDYE study: ABR NL 37479.042011). The aim of this study is to define the optimal dose of the fluorescent tracer Bevacizumab-IRDye800CW for intraoperative delineation of breast cancer tissue using the improved and optimized fluorescent tracer and camera system.

ELIGIBILITY:
Main Inclusion Criteria:

1. Females aged ≥ 18 years.
2. Confirmed diagnosis of breast cancer by means of histology or cytology and eligible for breast cancer surgery.
3. Tumor size ≥ 5 mm (0, 5 cm) diameter according to anatomical imaging data.
4. WHO performance score 0-2.
5. Life expectancy greater than 12 weeks
6. Written informed consent has been obtained
7. In the Investigator's opinion, patient is able and willing to comply with all trial requirements.

   For female subjects who are of childbearing potential, are premenopausal with intact reproductive organs or are less than 2 years post-menopausal:
8. A negative serum pregnancy test prior to receiving the second generation tracer
9. Willing to ensure that she or her partner uses effective contraception during the trial and for 3 months thereafter.

Main Exclusion Criteria:

1. Medical or psychiatric conditions that compromise the patient's ability to give informed consent
2. Breast prosthesis in the target breast
3. History of infusion reactions to Bevacizumab or other monoclonal antibody therapies
4. Concurrent anticancer therapy (chemotherapy, radiotherapy, vaccines, immunotherapy) delivered within the last 6 weeks prior to the start of the treatment
5. Significant renal or hepatic impairment.
6. Inadequately controlled hypertension with or without current antihypertensive medications.
7. History of myocardial infarction, transient ischemic attack, cerebro vascular accident, pulmonary embolism, uncontrolled congestive heart failure (CHF), significant liver disease, unstable angina within 6 months prior to enrollment.
8. Patients receiving anticoagulant therapy with vitamin K antagonists.
9. Patients receiving Class IA (e.g. Quinidine) or Class III (e.g. Dofetilide, Amiodarone, Sotalol) antiarrhythmic agents.
10. Evidence of QT prolongation on pre-treatment ECG (Males >440 ms, Females >450 ms).
11. Magnesium, potassium and calcium levels below lower normal limit which is regarded clinically relevant with regards to study participation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-10; Primary Completion 2017-01 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Tumor-to-background ratio | day 3

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events | up to two weeks

CONTACTS AND LOCATIONS:
Overall Officials: G.M van Dam, prof. dr., Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands